CLINICAL TRIAL: NCT06099912
Title: Individualized Dynamic Frailty-tailored Therapy (DynaFiT) in Elderly Patients With Newly Diagnosed Multiple Myeloma: a Prospective and Multi-center Study
Brief Title: Individualized Dynamic Frailty-tailored Therapy (DynaFiT) in Elderly Patients With NDMM
Acronym: DynaFiT
Status: Recruiting | Type: Observational
Sponsor: FengYan Jin (Other)
Collaborators: Sun Yat-sen University (Other); Ruijin Hospital (Other); Second Hospital of Shanxi Medical University (Other); The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Sponsor-Investigator, FengYan Jin, Clinical Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: DynaFiT
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Frailty
Keywords: Newly diagnosed multiple myeloma; Frailty; Elderly; Dynamic frailty-tailored therapy
MeSH Terms: conditions — Multiple Myeloma; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is dynamic and confers poor outcomes in elderly patients with newly diagnosed multiple myeloma (NDMM), mainly because of the high prevalence of treatment discontinuation due to intolerability. We designed a multi-center prospective study (DynaFiT) based on our real-life practice to evaluate the feasibility and benefits of a dynamic frailty-tailored therapy in elderly patients with different fitness/frailty statuses.

Since Dara-based treatment have recently become the new standard regimens, in this amendment of the study, daratumumab added to VRd is recommended as induction therapy regimen.

DETAILED DESCRIPTION:
Older patients with MM represent a heterogeneous population with different fitness/frailty statuses. Unlike fit patients who can benefit from intensive therapies due to their endurance, frail patients are often susceptible to treatment-related toxicity, leading to treatment discontinuation and poor outcomes. More importantly, frailty can diminish the prognostic impact of disease-related factors over disease trajectory. Thus, it is of utmost importance to determine the fitness/frailty status for treatment decision-making that carefully balances efficacy and safety in this vulnerable population. However, geriatric assessment is often conducted at diagnosis in clinical practice. Although baseline frailty status, as a static risk factor, is significantly associated with OS, its predictive ability decreases over time. Of note, emerging evidence indicates that the fitness/frailty status is highly dynamic because of age increase, disease trajectory, and treatment, raising the notion that frailty-tailored therapy should be designed based on the baseline fitness/frailty status and also according to its longitudinal changes during the treatment course. Thus, current frailty status better predicts OS.

To improve outcomes in elderly patients, this study was designed to investigate an entirely novel therapeutic strategy, the dynamic frailty-tailored therapy, in elderly MM patients with different fitness/frailty statuses.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged ≥65 years who were either transplant-ineligible or had no intent for immediate transplant;
* Subject must have documented multiple myeloma as defined by the criteria below:

Monoclonal plasma cells in the bone marrow 10% or presence of a biopsy-proven plasmacytoma;

Measurable disease as defined by any of the following:

* Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or
* IgA multiple myeloma: serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
* Light chain multiple myeloma: Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.

  * Has not had prior systemic therapy for multiple myeloma;
  * The functional reserve of the organs can withstand systemic therapy;
  * Each subject (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.

Exclusion Criteria:

* There are active systemic viral, fungal, or bacterial infections that require systemic anti-infective treatment;
* Severe organ dysfunction (New York Heart Association class III and IV or transaminases ≥5 normal level, except those caused by cardiac and hepatic amyloidosis secondary to MM)
* Patients with prior history of hematologic or solid tumors treated with radiotherapy or chemotherapy(except ≥5 years);
* Patients who currently have hematologic tumors or solid tumors that require radiotherapy or chemotherapy;
* Non-signation of informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Diagnosed with primary multiple myeloma according to the 2014 IMWG multiple myeloma diagnostic criteria,aged ≥65 years who were either transplant-ineligible or had no intent for immediate transplant.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2029-09-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (at least PR) on induction therapy | From the date of inclusion to the end of induction therapy, up to 8 months.
  Overall response rate(ORR) is defined as the percentage of participants with presence of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). ORR assessment will be based on International Myeloma Working Group (IMWG) response criteria.

SECONDARY OUTCOMES:
Rate of treatment discontinued(TD) | The time from the date of inclusion to the date of treatment discontinued from any cause, up to 24 months.
  The effect of intensive or mild treatment based on dynamic frailty status on treatment discontinued(TD) in elderly newly diagnosed multiple myeloma.
Treatment related adverse event(TRAE) | Baseline, end of every induction cycle and maintenance cycle, until disease progression or treatment discontinued, up to 24 months.
  Toxicity and safety will be reported based on the adverse events, as graded by CTCAE V5 and determined by routine clinical assessments.
Early mortality(EM) | The time from the date of inclusion to the date of death from any cause, up to 24 months.
  Early mortality is defined as death within 3, 6, 12 and 24 months (EM3,EM6,EM12 and EM24).
Progression-free survival(PFS) | The time from the date of inclusion to the date of first documented evidence of disease progression or death from any cause, up to 24 months.
  Progression-free survival(PFS) is defined as the time from inclusion to the time of first documented evidence of disease progression or death from any cause. Individuals who are lost to follow-up or progression-free at the time of analysis will be censored at their last known date to be alive and progression-free. Disease progression is defined according to the IMWG Uniform Response Criteria for Multiple Myeloma.
Overall survival (OS) | The time from the date of inclusion to the date of death from any cause, up to 24 months
  In each case it is the time from inclusion to the time of death from any cause. Individuals who are lost to follow-up or still alive at the time of analysis will be censored at their last known date to be alive.

OTHER OUTCOMES:
To establish a new and better comprehensive geriatric assessment system to predict prognosis of elderly NDMM | Through study completion, up to 24 months.
  To establish a new and better comprehensive geriatric frailty assessment system that can predict TD and OS in NDMM patients, combining objective biological markers (biomarkers of sarcopenia, n-terminal pro-brain natriuretic peptide, inflammatory markers such as C-reactive protein, aging biomarkers, and immune markers).
To explore the value of sarcopenia in predicting treatment discontinued(TD) and prognosis of the elderly newly diagnosed multiple myeloma | Through study completion, up to 24 months.
  Number of participants with imaging sarcopenia as assessed by dual-energy X-ray absorptiometry and whole-body low-dose CT;Number of participants with functional sarcopenia as assessed by grip strength and 6-meter walking speed;Number of participants with objective biomarkers in sarcopenia as assessed by peripheral blood test.
Minimal residual disease (MRD) | Through study completion, up to 24 months.
  By using multiparameter flow cytometry and/or next-generation sequencing techniques dynamically monitor MRD status and its effect on OS and PFS
Discovery and identification of frailty biomarkers in elderly newly diagnosed multiple myeloma | Through study completion, up to 24 months.
  Discovery and identification of frailty biomarkers in elderly newly diagnosed multiple myeloma.
To explore the prognostic significance of blood liquid biopsy based on platelet RNA sequencing for multiple myeloma | Through study completion, up to 24 months.
  Heterogeneity of disease as assessed by platelet RNA sequencing to explore the prognostic significance of blood liquid biopsy based on for multiple myeloma.
To establish a predictive model for treatment discontinuation in elderly NDMM. | The time from the date of inclusion to the date of treatment discontinued, up to 24 months
  To identify elderly NDMM who are intolerant to standard-dose therapy, a predictive model for treatment discontinuation will be constructed. Proactive management will be implemented for patients at high risk of treatment discontinuation, including appropriate reduction of treatment intensity and active supportive care.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar SK, Rajkumar V, Kyle RA, van Duin M, Sonneveld P, Mateos MV, Gay F, Anderson KC. Multiple myeloma. Nat Rev Dis Primers. 2017 Jul 20;3:17046. doi: 10.1038/nrdp.2017.46. PMID 28726797
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Abate D, Abbasi N, Abbastabar H, Abd-Allah F, Abdel-Rahman O, Abdelalim A, Abdoli A, Abdollahpour I, Abdulle ASM, Abebe ND, Abraha HN, Abu-Raddad LJ, Abualhasan A, Adedeji IA, Advani SM, Afarideh M, Afshari M, Aghaali M, Agius D, Agrawal S, Ahmadi A, Ahmadian E, Ahmadpour E, Ahmed MB, Akbari ME, Akinyemiju T, Al-Aly Z, AlAbdulKader AM, Alahdab F, Alam T, Alamene GM, Alemnew BTT, Alene KA, Alinia C, Alipour V, Aljunid SM, Bakeshei FA, Almadi MAH, Almasi-Hashiani A, Alsharif U, Alsowaidi S, Alvis-Guzman N, Amini E, Amini S, Amoako YA, Anbari Z, Anber NH, Andrei CL, Anjomshoa M, Ansari F, Ansariadi A, Appiah SCY, Arab-Zozani M, Arabloo J, Arefi Z, Aremu O, Areri HA, Artaman A, Asayesh H, Asfaw ET, Ashagre AF, Assadi R, Ataeinia B, Atalay HT, Ataro Z, Atique S, Ausloos M, Avila-Burgos L, Avokpaho EFGA, Awasthi A, Awoke N, Ayala Quintanilla BP, Ayanore MA, Ayele HT, Babaee E, Bacha U, Badawi A, Bagherzadeh M, Bagli E, Balakrishnan S, Balouchi A, Barnighausen TW, Battista RJ, Behzadifar M, Behzadifar M, Bekele BB, Belay YB, Belayneh YM, Berfield KKS, Berhane A, Bernabe E, Beuran M, Bhakta N, Bhattacharyya K, Biadgo B, Bijani A, Bin Sayeed MS, Birungi C, Bisignano C, Bitew H, Bjorge T, Bleyer A, Bogale KA, Bojia HA, Borzi AM, Bosetti C, Bou-Orm IR, Brenner H, Brewer JD, Briko AN, Briko NI, Bustamante-Teixeira MT, Butt ZA, Carreras G, Carrero JJ, Carvalho F, Castro C, Castro F, Catala-Lopez F, Cerin E, Chaiah Y, Chanie WF, Chattu VK, Chaturvedi P, Chauhan NS, Chehrazi M, Chiang PP, Chichiabellu TY, Chido-Amajuoyi OG, Chimed-Ochir O, Choi JJ, Christopher DJ, Chu DT, Constantin MM, Costa VM, Crocetti E, Crowe CS, Curado MP, Dahlawi SMA, Damiani G, Darwish AH, Daryani A, das Neves J, Demeke FM, Demis AB, Demissie BW, Demoz GT, Denova-Gutierrez E, Derakhshani A, Deribe KS, Desai R, Desalegn BB, Desta M, Dey S, Dharmaratne SD, Dhimal M, Diaz D, Dinberu MTT, Djalalinia S, Doku DT, Drake TM, Dubey M, Dubljanin E, Duken EE, Ebrahimi H, Effiong A, Eftekhari A, El Sayed I, Zaki MES, El-Jaafary SI, El-Khatib Z, Elemineh DA, Elkout H, Ellenbogen RG, Elsharkawy A, Emamian MH, Endalew DA, Endries AY, Eshrati B, Fadhil I, Fallah Omrani V, Faramarzi M, Farhangi MA, Farioli A, Farzadfar F, Fentahun N, Fernandes E, Feyissa GT, Filip I, Fischer F, Fisher JL, Force LM, Foroutan M, Freitas M, Fukumoto T, Futran ND, Gallus S, Gankpe FG, Gayesa RT, Gebrehiwot TT, Gebremeskel GG, Gedefaw GA, Gelaw BK, Geta B, Getachew S, Gezae KE, Ghafourifard M, Ghajar A, Ghashghaee A, Gholamian A, Gill PS, Ginindza TTG, Girmay A, Gizaw M, Gomez RS, Gopalani SV, Gorini G, Goulart BNG, Grada A, Ribeiro Guerra M, Guimaraes ALS, Gupta PC, Gupta R, Hadkhale K, Haj-Mirzaian A, Haj-Mirzaian A, Hamadeh RR, Hamidi S, Hanfore LK, Haro JM, Hasankhani M, Hasanzadeh A, Hassen HY, Hay RJ, Hay SI, Henok A, Henry NJ, Herteliu C, Hidru HD, Hoang CL, Hole MK, Hoogar P, Horita N, Hosgood HD, Hosseini M, Hosseinzadeh M, Hostiuc M, Hostiuc S, Househ M, Hussen MM, Ileanu B, Ilic MD, Innos K, Irvani SSN, Iseh KR, Islam SMS, Islami F, Jafari Balalami N, Jafarinia M, Jahangiry L, Jahani MA, Jahanmehr N, Jakovljevic M, James SL, Javanbakht M, Jayaraman S, Jee SH, Jenabi E, Jha RP, Jonas JB, Jonnagaddala J, Joo T, Jungari SB, Jurisson M, Kabir A, Kamangar F, Karch A, Karimi N, Karimian A, Kasaeian A, Kasahun GG, Kassa B, Kassa TD, Kassaw MW, Kaul A, Keiyoro PN, Kelbore AG, Kerbo AA, Khader YS, Khalilarjmandi M, Khan EA, Khan G, Khang YH, Khatab K, Khater A, Khayamzadeh M, Khazaee-Pool M, Khazaei S, Khoja AT, Khosravi MH, Khubchandani J, Kianipour N, Kim D, Kim YJ, Kisa A, Kisa S, Kissimova-Skarbek K, Komaki H, Koyanagi A, Krohn KJ, Bicer BK, Kugbey N, Kumar V, Kuupiel D, La Vecchia C, Lad DP, Lake EA, Lakew AM, Lal DK, Lami FH, Lan Q, Lasrado S, Lauriola P, Lazarus JV, Leigh J, Leshargie CT, Liao Y, Limenih MA, Listl S, Lopez AD, Lopukhov PD, Lunevicius R, Madadin M, Magdeldin S, El Razek HMA, Majeed A, Maleki A, Malekzadeh R, Manafi A, Manafi N, Manamo WA, Mansourian M, Mansournia MA, Mantovani LG, Maroufizadeh S, Martini SMS, Mashamba-Thompson TP, Massenburg BB, Maswabi MT, Mathur MR, McAlinden C, McKee M, Meheretu HAA, Mehrotra R, Mehta V, Meier T, Melaku YA, Meles GG, Meles HG, Melese A, Melku M, Memiah PTN, Mendoza W, Menezes RG, Merat S, Meretoja TJ, Mestrovic T, Miazgowski B, Miazgowski T, Mihretie KMM, Miller TR, Mills EJ, Mir SM, Mirzaei H, Mirzaei HR, Mishra R, Moazen B, Mohammad DK, Mohammad KA, Mohammad Y, Darwesh AM, Mohammadbeigi A, Mohammadi H, Mohammadi M, Mohammadian M, Mohammadian-Hafshejani A, Mohammadoo-Khorasani M, Mohammadpourhodki R, Mohammed AS, Mohammed JA, Mohammed S, Mohebi F, Mokdad AH, Monasta L, Moodley Y, Moosazadeh M, Moossavi M, Moradi G, Moradi-Joo M, Moradi-Lakeh M, Moradpour F, Morawska L, Morgado-da-Costa J, Morisaki N, Morrison SD, Mosapour A, Mousavi SM, Muche AA, Muhammed OSS, Musa J, Nabhan AF, Naderi M, Nagarajan AJ, Nagel G, Nahvijou A, Naik G, Najafi F, Naldi L, Nam HS, Nasiri N, Nazari J, Negoi I, Neupane S, Newcomb PA, Nggada HA, Ngunjiri JW, Nguyen CT, Nikniaz L, Ningrum DNA, Nirayo YL, Nixon MR, Nnaji CA, Nojomi M, Nosratnejad S, Shiadeh MN, Obsa MS, Ofori-Asenso R, Ogbo FA, Oh IH, Olagunju AT, Olagunju TO, Oluwasanu MM, Omonisi AE, Onwujekwe OE, Oommen AM, Oren E, Ortega-Altamirano DDV, Ota E, Otstavnov SS, Owolabi MO, P A M, Padubidri JR, Pakhale S, Pakpour AH, Pana A, Park EK, Parsian H, Pashaei T, Patel S, Patil ST, Pennini A, Pereira DM, Piccinelli C, Pillay JD, Pirestani M, Pishgar F, Postma MJ, Pourjafar H, Pourmalek F, Pourshams A, Prakash S, Prasad N, Qorbani M, Rabiee M, Rabiee N, Radfar A, Rafiei A, Rahim F, Rahimi M, Rahman MA, Rajati F, Rana SM, Raoofi S, Rath GK, Rawaf DL, Rawaf S, Reiner RC, Renzaho AMN, Rezaei N, Rezapour A, Ribeiro AI, Ribeiro D, Ronfani L, Roro EM, Roshandel G, Rostami A, Saad RS, Sabbagh P, Sabour S, Saddik B, Safiri S, Sahebkar A, Salahshoor MR, Salehi F, Salem H, Salem MR, Salimzadeh H, Salomon JA, Samy AM, Sanabria J, Santric Milicevic MM, Sartorius B, Sarveazad A, Sathian B, Satpathy M, Savic M, Sawhney M, Sayyah M, Schneider IJC, Schottker B, Sekerija M, Sepanlou SG, Sepehrimanesh M, Seyedmousavi S, Shaahmadi F, Shabaninejad H, Shahbaz M, Shaikh MA, Shamshirian A, Shamsizadeh M, Sharafi H, Sharafi Z, Sharif M, Sharifi A, Sharifi H, Sharma R, Sheikh A, Shirkoohi R, Shukla SR, Si S, Siabani S, Silva DAS, Silveira DGA, Singh A, Singh JA, Sisay S, Sitas F, Sobngwi E, Soofi M, Soriano JB, Stathopoulou V, Sufiyan MB, Tabares-Seisdedos R, Tabuchi T, Takahashi K, Tamtaji OR, Tarawneh MR, Tassew SG, Taymoori P, Tehrani-Banihashemi A, Temsah MH, Temsah O, Tesfay BE, Tesfay FH, Teshale MY, Tessema GA, Thapa S, Tlaye KG, Topor-Madry R, Tovani-Palone MR, Traini E, Tran BX, Tran KB, Tsadik AG, Ullah I, Uthman OA, Vacante M, Vaezi M, Varona Perez P, Veisani Y, Vidale S, Violante FS, Vlassov V, Vollset SE, Vos T, Vosoughi K, Vu GT, Vujcic IS, Wabinga H, Wachamo TM, Wagnew FS, Waheed Y, Weldegebreal F, Weldesamuel GT, Wijeratne T, Wondafrash DZ, Wonde TE, Wondmieneh AB, Workie HM, Yadav R, Yadegar A, Yadollahpour A, Yaseri M, Yazdi-Feyzabadi V, Yeshaneh A, Yimam MA, Yimer EM, Yisma E, Yonemoto N, Younis MZ, Yousefi B, Yousefifard M, Yu C, Zabeh E, Zadnik V, Moghadam TZ, Zaidi Z, Zamani M, Zandian H, Zangeneh A, Zaki L, Zendehdel K, Zenebe ZM, Zewale TA, Ziapour A, Zodpey S, Murray CJL. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2017: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2019 Dec 1;5(12):1749-1768. doi: 10.1001/jamaoncol.2019.2996. PMID 31560378
- [Background] Kumar SK, Dispenzieri A, Lacy MQ, Gertz MA, Buadi FK, Pandey S, Kapoor P, Dingli D, Hayman SR, Leung N, Lust J, McCurdy A, Russell SJ, Zeldenrust SR, Kyle RA, Rajkumar SV. Continued improvement in survival in multiple myeloma: changes in early mortality and outcomes in older patients. Leukemia. 2014 May;28(5):1122-8. doi: 10.1038/leu.2013.313. Epub 2013 Oct 25. PMID 24157580
- [Background] Cardoso AL, Fernandes A, Aguilar-Pimentel JA, de Angelis MH, Guedes JR, Brito MA, Ortolano S, Pani G, Athanasopoulou S, Gonos ES, Schosserer M, Grillari J, Peterson P, Tuna BG, Dogan S, Meyer A, van Os R, Trendelenburg AU. Towards frailty biomarkers: Candidates from genes and pathways regulated in aging and age-related diseases. Ageing Res Rev. 2018 Nov;47:214-277. doi: 10.1016/j.arr.2018.07.004. Epub 2018 Jul 30. PMID 30071357
- [Background] Bringhen S, Mateos MV, Zweegman S, Larocca A, Falcone AP, Oriol A, Rossi D, Cavalli M, Wijermans P, Ria R, Offidani M, Lahuerta JJ, Liberati AM, Mina R, Callea V, Schaafsma M, Cerrato C, Marasca R, Franceschini L, Evangelista A, Teruel AI, van der Holt B, Montefusco V, Ciccone G, Boccadoro M, San Miguel J, Sonneveld P, Palumbo A. Age and organ damage correlate with poor survival in myeloma patients: meta-analysis of 1435 individual patient data from 4 randomized trials. Haematologica. 2013 Jun;98(6):980-7. doi: 10.3324/haematol.2012.075051. Epub 2013 Feb 26. PMID 23445873
- [Background] Palumbo A, Avet-Loiseau H, Oliva S, Lokhorst HM, Goldschmidt H, Rosinol L, Richardson P, Caltagirone S, Lahuerta JJ, Facon T, Bringhen S, Gay F, Attal M, Passera R, Spencer A, Offidani M, Kumar S, Musto P, Lonial S, Petrucci MT, Orlowski RZ, Zamagni E, Morgan G, Dimopoulos MA, Durie BG, Anderson KC, Sonneveld P, San Miguel J, Cavo M, Rajkumar SV, Moreau P. Revised International Staging System for Multiple Myeloma: A Report From International Myeloma Working Group. J Clin Oncol. 2015 Sep 10;33(26):2863-9. doi: 10.1200/JCO.2015.61.2267. Epub 2015 Aug 3. PMID 26240224
- [Background] Palumbo A, Bringhen S, Mateos MV, Larocca A, Facon T, Kumar SK, Offidani M, McCarthy P, Evangelista A, Lonial S, Zweegman S, Musto P, Terpos E, Belch A, Hajek R, Ludwig H, Stewart AK, Moreau P, Anderson K, Einsele H, Durie BG, Dimopoulos MA, Landgren O, San Miguel JF, Richardson P, Sonneveld P, Rajkumar SV. Geriatric assessment predicts survival and toxicities in elderly myeloma patients: an International Myeloma Working Group report. Blood. 2015 Mar 26;125(13):2068-74. doi: 10.1182/blood-2014-12-615187. Epub 2015 Jan 27. PMID 25628469
- [Background] Coulson AB, Royle KL, Pawlyn C, Cairns DA, Hockaday A, Bird J, Bowcock S, Kaiser M, de Tute R, Rabin N, Boyd K, Jones J, Parrish C, Gardner H, Meads D, Dawkins B, Olivier C, Henderson R, Best P, Owen R, Jenner M, Kishore B, Drayson M, Jackson G, Cook G. Frailty-adjusted therapy in Transplant Non-Eligible patients with newly diagnosed Multiple Myeloma (FiTNEss (UK-MRA Myeloma XIV Trial)): a study protocol for a randomised phase III trial. BMJ Open. 2022 Jun 2;12(6):e056147. doi: 10.1136/bmjopen-2021-056147. PMID 35654466
- [Background] Yao Y, Sui WW, Liao AJ, Wang W, Chen LJ, Chu XX, Bao L, Cen XN, Fu R, Liu H, Sun CY, Jin FY, Yan H, Wang LQ, Yuan CL, Gao GX, Gao D, Zhang JQ, He JX, Hu JD, Ma LM, Zhang L, Zhou DB, Zou DH, Li J. Comprehensive geriatric assessment in newly diagnosed older myeloma patients: a multicentre, prospective, non-interventional study. Age Ageing. 2022 Jan 6;51(1):afab211. doi: 10.1093/ageing/afab211. PMID 34673897
- [Background] Larocca A, Dold SM, Zweegman S, Terpos E, Wasch R, D'Agostino M, Scheubeck S, Goldschmidt H, Gay F, Cavo M, Ludwig H, Straka C, Bringhen S, Auner HW, Caers J, Gramatzki M, Offidani M, Dimopoulos MA, Einsele H, Boccadoro M, Sonneveld P, Engelhardt M. Patient-centered practice in elderly myeloma patients: an overview and consensus from the European Myeloma Network (EMN). Leukemia. 2018 Aug;32(8):1697-1712. doi: 10.1038/s41375-018-0142-9. Epub 2018 Apr 25. PMID 29880892
- [Background] Stege CAM, Nasserinejad K, van der Spek E, Bilgin YM, Kentos A, Sohne M, van Kampen RJW, Ludwig I, Thielen N, Durdu-Rayman N, de Graauw NCHP, van de Donk NWCJ, de Waal EGM, Vekemans MC, Timmers GJ, van der Klift M, Soechit S, Geerts PAF, Silbermann MH, Oosterveld M, Nijhof IS, Sonneveld P, Klein SK, Levin MD, Zweegman S. Ixazomib, Daratumumab, and Low-Dose Dexamethasone in Frail Patients With Newly Diagnosed Multiple Myeloma: The Hovon 143 Study. J Clin Oncol. 2021 Sep 1;39(25):2758-2767. doi: 10.1200/JCO.20.03143. Epub 2021 May 4. PMID 33945289
- [Background] Stege CAM, Nasserinejad K, Klein SK, Timmers GJ, Hoogendoorn M, Ypma PF, Nijhof IS, Velders GA, Strobbe L, Durdu-Rayman N, Westerman M, Davidis-van Schoonhoven MA, van Kampen RJW, Beeker A, Koster A, Dijk AC, van de Donk NWCJ, van der Spek E, Leys RBL, Silbermann MH, Groen K, van der Burg-de Graauw NCHP, Sinnige HAM, van der Hem KG, Levenga H, Bilgin YM, Sonneveld P, Levin MD, Zweegman S. Improving the identification of frail elderly newly diagnosed multiple myeloma patients. Leukemia. 2021 Sep;35(9):2715-2719. doi: 10.1038/s41375-021-01162-z. Epub 2021 Feb 15. No abstract available. PMID 33589752
- [Background] Antoine-Pepeljugoski C, Braunstein MJ. Management of Newly Diagnosed Elderly Multiple Myeloma Patients. Curr Oncol Rep. 2019 May 24;21(7):64. doi: 10.1007/s11912-019-0804-4. PMID 31127403
- [Background] Mina R, Bringhen S, Wildes TM, Zweegman S, Rosko AE. Approach to the Older Adult With Multiple Myeloma. Am Soc Clin Oncol Educ Book. 2019 Jan;39:500-518. doi: 10.1200/EDBK_239067. Epub 2019 May 17. PMID 31099676
- [Background] Joao C, Geraldes C, Neves M, Mariz M, Trigo F. Management of older and frail patients with multiple myeloma in the Portuguese routine clinical practice: Deliberations and recommendations from an expert panel of hematologists. J Geriatr Oncol. 2020 Nov;11(8):1210-1216. doi: 10.1016/j.jgo.2020.06.002. Epub 2020 Jun 27. PMID 32601004
- [Background] Mian H, Wildes TM, Vij R, Pianko MJ, Major A, Fiala MA. Dynamic frailty risk assessment among older adults with multiple myeloma: A population-based cohort study. Blood Cancer J. 2023 May 10;13(1):76. doi: 10.1038/s41408-023-00843-5. PMID 37164972
- [Background] Raje NS, Anaissie E, Kumar SK, Lonial S, Martin T, Gertz MA, Krishnan A, Hari P, Ludwig H, O'Donnell E, Yee A, Kaufman JL, Cohen AD, Garderet L, Wechalekar AF, Terpos E, Khatry N, Niesvizky R, Yi Q, Joshua DE, Saikia T, Leung N, Engelhardt M, Mothy M, Branagan A, Chari A, Reiman AJ, Lipe B, Richter J, Rajkumar SV, Miguel JS, Anderson KC, Stadtmauer EA, Prabhala RH, McCarthy PL, Munshi NC. Consensus guidelines and recommendations for infection prevention in multiple myeloma: a report from the International Myeloma Working Group. Lancet Haematol. 2022 Feb;9(2):e143-e161. doi: 10.1016/S2352-3026(21)00283-0. PMID 35114152
- [Background] Encinas C, Hernandez-Rivas JA, Oriol A, Rosinol L, Blanchard MJ, Bellon JM, Garcia-Sanz R, de la Rubia J, de la Guia AL, Jimenez-Ubieto A, Jarque I, Inigo B, Dourdil V, de Arriba F, Perez-Avila CC, Gonzalez Y, Hernandez MT, Bargay J, Granell M, Rodriguez-Otero P, Silvent M, Cabrera C, Rios R, Alegre A, Gironella M, Gonzalez MS, Sureda A, Sampol A, Ocio EM, Krsnik I, Garcia A, Garcia-Mateo A, Soler JA, Martin J, Arguinano JM, Mateos MV, Blade J, San-Miguel JF, Lahuerta JJ, Martinez-Lopez J; GEM/PETHEMA (Grupo Espanol de Mieloma/Programa para el Estudio de la Terapeutica en Hemopatias Malignas) cooperative study group. A simple score to predict early severe infections in patients with newly diagnosed multiple myeloma. Blood Cancer J. 2022 Apr 19;12(4):68. doi: 10.1038/s41408-022-00652-2. PMID 35440057
- [Derived] Zhang Y, Liang X, Xu W, Yi X, Hu R, Ma X, Yan Y, Zhang N, Wang J, Sun X, Zhu Y, Tian M, Lan M, Long M, Dai Y, Jin F. Individualized dynamic frailty-tailored therapy (DynaFiT) in elderly patients with newly diagnosed multiple myeloma: a prospective study. J Hematol Oncol. 2024 Jun 24;17(1):48. doi: 10.1186/s13045-024-01569-y. PMID 38915117